CLINICAL TRIAL: NCT00364338
Title: Development of Gourmet Medical Cooking Workshop for Lifestyle Changing and Its Affect on Perimenopausal Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 30-150906-HMO-CTIL
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2006-08

CONDITIONS: Perimenopausal
Keywords: gourmet healthy cooking; quality of life; preimenopause; weight; lipids
MeSH Terms: conditions — Body Weight

INTERVENTIONS:
Behavioral: gourment cooking workshop

SUMMARY:
Subjects that participate in the practical workshop will improve their metabolic indexes, decrease their weight and improve their quality of life, in contrast to the participants that will take part in the nutritional consulting sessions

DETAILED DESCRIPTION:
Participants will be randomly assigned to a dietary consultation-only control group or to a gourmet medical cooking workshop. The workshop will consist of 9 lessons with the following lessons: introduction, fats, phytoestrogens, carbohydrates and fibers, calcium and low calorie diet, party's recipes, shopping and farewell dinner. All the lessons will start with half an hour theoretical introduction, followed by a 2.5 hours "hands on" session under supervision of a medical chef. The study population will include healthy women attending the menopause clinic. 72 patients will be recruited and will be randomly divided into two groups: an intervention group of 36 will commence the workshop during 2007 and a control group of 36 who will take part in dietitian consulting sessions only. During 2008 the control group will commence the workshop and will add to the study group.

ELIGIBILITY:
Inclusion Criteria:

* Age of 45-60
* Perimenopause
* Healthy
* BMI over 17

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
We expect to see change in the following outcomes:
the patient's metabolic state,
the patient's weight
body composite
patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: ronit kochman, md, Principal Investigator — hadassah university hospital
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel